CLINICAL TRIAL: NCT04620993
Title: Investigation of the Effect of Biomechanical and Viscoelastic Properties of Plantar Fascia on Pelvic Girdle Pain in Pregnant Women
Brief Title: Biomechanical and Viscoelastic Properties of Plantar Fascia in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 166
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2020-11

CONDITIONS: Pelvic Girdle Pain; Biomechanical and Viscoelastic Properties of Plantar Fascia; Pregnant Woman
Keywords: pelvic girdle pain, pregnant women, plantar fascia
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: pregnant women with pelvic girdle pain: This group will consist of pregnant women who are in the 2nd or 3rd trimester of pregnancy and have pelvic girdle pain.
  Interventions: Other: Evaluation of biomechanics and viscoelastic properties of plantar fascia; Other: Evaluation of navıcular drop; Other: Evaluation of plantar pressure distrubution
- Group 2:pregnant women without pelvic girdle pain: This group will consist of pregnant women who are in the 2nd or 3rd trimester of pregnancy but have not pelvic girdle pain.
  Interventions: Other: Evaluation of biomechanics and viscoelastic properties of plantar fascia; Other: Evaluation of navıcular drop; Other: Evaluation of plantar pressure distrubution
- Group 3: healthy women: This group will consist of healthy women who have not been pregnant.
  Interventions: Other: Evaluation of biomechanics and viscoelastic properties of plantar fascia; Other: Evaluation of navıcular drop; Other: Evaluation of plantar pressure distrubution

INTERVENTIONS:
Other: Evaluation of biomechanics and viscoelastic properties of plantar fascia — The biomechanical and viscoelastic properties of the plantar fascia will be measured in the side lying position.
  Measurements will be made with the ankle in neutral position and maximum dorsi flexion position.
Other: Evaluation of navıcular drop — The amount of navicular drop of both feet will be measured
Other: Evaluation of plantar pressure distrubution — The distribution of foot plantar pressure and the amount of change in the center of gravity will be measured in the free standing position.

SUMMARY:
Pelvic girdle pain is frequently experienced in pregnant women and the mechanism of pelvic girdle pain is not known exactly. The aim of this study is to investigate the effect of biomechanical and viscoelastic properties of plantar fascia on pelvic girdle pain in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the 2nd or 3rd trimester of pregnancy with pelvic girdle pain
* Pregnant women in the 2nd or 3rd trimester of pregnancy without pelvic girdle pain
* First pregnancy
* 20-40 years old
* Healthy woman without pregnancy

Exclusion Criteria:

* Participant having any kind of connective tissue disease
* Presence of orthopedic or neurological problems in the lower extremities that may cause musculoskeletal disorder and biomechanical alignment deviations
* Presence of foot pain that started before pregnancy and lasts for more than 3 months
* Presence of lumbar-pelvic pain that started before pregnancy and lasts for more than 3 months
* Have had 2 or more births
* Presence of multiple pregnancy (twins, triplets etc)
* Presence of ankle-ankle fracture and operation history in the last 6 months

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pegnant women with pelvic girdle pain Pegnant women without pelvic girdle pain Non pregnant healthy women
Study Population: Pegnant women with pelvic girdle pain Pegnant women without pelvic girdle pain Non pregnant healthy women
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of biomechanical and viscoelastic properties of plantar fascia | Baseline Measurements
  Measuring of the biomechanical and viscoelastic properties of the plantar fascia (with MyotonPro, Myoton AS, Tallin, Estonia) in the side lying position.
Evaluation of plantar pressure distrubution | Baseline Measurements
  Measuring of plantar pressure distrubution (with Tekscan, Boston, MA, USA) in free standing position

SECONDARY OUTCOMES:
Evaluation of navicular drop | Baseline Measurements
  Measuring of the amount of the navicular drop

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Saglık Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Park SY, Park DJ. Comparison of Foot Structure, Function, Plantar Pressure and Balance Ability According to the Body Mass Index of Young Adults. Osong Public Health Res Perspect. 2019 Apr;10(2):102-107. doi: 10.24171/j.phrp.2019.10.2.09. PMID 31065537
- [Result] Elden H, Gutke A, Kjellby-Wendt G, Fagevik-Olsen M, Ostgaard HC. Predictors and consequences of long-term pregnancy-related pelvic girdle pain: a longitudinal follow-up study. BMC Musculoskelet Disord. 2016 Jul 12;17:276. doi: 10.1186/s12891-016-1154-0. PMID 27406174
- [Result] Bertuit J, Van Lint CE, Rooze M, Feipel V. Pregnancy and pelvic girdle pain: Analysis of pelvic belt on pain. J Clin Nurs. 2018 Jan;27(1-2):e129-e137. doi: 10.1111/jocn.13888. Epub 2017 Nov 3. PMID 28544276
- [Result] Kerbourc'h F, Bertuit J, Feipel V, Rooze M. Pregnancy and Pelvic Girdle PainAnalysis of Center of Pressure During Gait. J Am Podiatr Med Assoc. 2017 Jul;107(4):299-306. doi: 10.7547/15-087. PMID 28880594
- [Result] Aldabe D, Ribeiro DC, Milosavljevic S, Dawn Bussey M. Pregnancy-related pelvic girdle pain and its relationship with relaxin levels during pregnancy: a systematic review. Eur Spine J. 2012 Sep;21(9):1769-76. doi: 10.1007/s00586-012-2162-x. Epub 2012 Feb 4. PMID 22310881
- [Result] Ceprnja D, Chipchase L, Gupta A. Prevalence of pregnancy-related pelvic girdle pain and associated factors in Australia: a cross-sectional study protocol. BMJ Open. 2017 Nov 15;7(11):e018334. doi: 10.1136/bmjopen-2017-018334. PMID 29146651
- [Result] Wuytack F, Daly D, Curtis E, Begley C. Prognostic factors for pregnancy-related pelvic girdle pain, a systematic review. Midwifery. 2018 Nov;66:70-78. doi: 10.1016/j.midw.2018.07.012. Epub 2018 Aug 8. PMID 30142609
- [Result] Aldabe D, Milosavljevic S, Bussey MD. Is pregnancy related pelvic girdle pain associated with altered kinematic, kinetic and motor control of the pelvis? A systematic review. Eur Spine J. 2012 Sep;21(9):1777-87. doi: 10.1007/s00586-012-2401-1. Epub 2012 Jun 21. PMID 22718046
- [Result] Khamis S, Yizhar Z. Effect of feet hyperpronation on pelvic alignment in a standing position. Gait Posture. 2007 Jan;25(1):127-34. doi: 10.1016/j.gaitpost.2006.02.005. Epub 2006 Apr 18. PMID 16621569